CLINICAL TRIAL: NCT07173439
Title: A Multi-center, Prospective, Single Blinded, Randomized, Comparative, Pivotal Clinical Trial to Evaluate the Efficacy and Safety of Digital Therapeutics to Improve ADHD Symptoms of Patients Diagnosed With ADHD
Brief Title: Multi-center, Single Blinded, RCT, Pivotal Study to Evaluate the Efficacy and Safety of DTx to Improve ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EMOTIV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EM_SNU_001
Record Dates: First submitted 2025-08-20; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; ADHD - Combined Type; ADHD
Keywords: ADHD; DTx
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The treatment group used the device with driving and N-BACK cognitive training functions. (Experimental): The treatment group participated in the clinical trial by using the investigational digital therapeutic device, which incorporated both driving simulation and N-BACK cognitive training functions. These features were designed to engage and improve key cognitive abilities such as attention, working memory, and executive function, which are often impaired in individuals with ADHD. The combined use of driving tasks and N-BACK exercises aimed to provide a comprehensive and interactive therapeutic intervention to help reduce core ADHD symptoms.
  Interventions: Device: Model Name: EMT-SR01;red
- The control group used a device that included only the driving function, without the N-BACK cognitiv (Sham Comparator): The control group participated in the clinical trial using a digital device that incorporated only the driving simulation function. Unlike the treatment group, this device did not include the N-BACK cognitive training component. The driving function served as a digital placebo (sham) intervention designed to mimic the user experience without providing the active therapeutic elements targeting cognitive functions. This setup allowed for a controlled comparison to evaluate the efficacy of the combined intervention in the treatment group.
  Interventions: Device: Model Name: EMT-SR01;red (Placebo)

INTERVENTIONS:
Device: Model Name: EMT-SR01;red — The investigational device incorporated both a driving simulation and an N-Back cognitive training function. These features were designed to engage and improve key cognitive abilities such as attention, working memory, and executive function, which are often impaired in individuals with ADHD. The combined use of driving tasks and N-Back exercises aimed to provide a comprehensive and interactive therapeutic intervention to reduce core ADHD symptoms.
  Arms: The treatment group used the device with driving and N-BACK cognitive training functions.
Device: Model Name: EMT-SR01;red (Placebo) — The placebo device incorporated only the driving simulation function and excluded the N-Back cognitive training component. The driving simulation was designed as a sham intervention to mimic the user experience without providing the active therapeutic elements targeting cognitive functions. This setup enabled a controlled comparison with the active digital therapeutic device.
  Arms: The control group used a device that included only the driving function, without the N-BACK cognitiv

SUMMARY:
Background:

Attention Deficit Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by inattention, hyperactivity, impulsivity, and impaired executive functioning. It typically begins in childhood and is often first diagnosed at school age due to learning and social behavioral difficulties. Therefore, ADHD treatment aims to directly enhance attention, reduce hyperactivity and impulsivity, and ultimately improve task performance and associated behavioral and relational issues.

Objective of the Clinical Trial:

To evaluate the safety of the investigational digital therapeutic device for the treatment of ADHD.

To evaluate the efficacy of the investigational digital therapeutic device for the treatment of ADHD.

Study Design & Methodology:

A total of 122 participants were enrolled (62 in the treatment group and 60 in the control group), with 114 participants included in the Full Analysis Set (FAS: 58 treatment, 56 control).

DETAILED DESCRIPTION:
Expanded Clinical Summary: Investigational Digital Therapeutic Device for ADHD

[Background and Rationale] Attention-Deficit/Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder characterized by a persistent pattern of inattention, hyperactivity, impulsivity, and impairments in executive function. These symptoms typically begin in childhood and are often first identified in school-aged children due to learning difficulties or social behavioral issues.

Effective treatment of ADHD aims to improve sustained attention, reduce hyperactivity and impulsivity, and enhance the patient's ability to engage in academic, social, and daily life activities. While pharmacological interventions have been the mainstay of treatment, increasing attention has been directed toward non-pharmacologic and digital therapeutic approaches, particularly those that can target cognitive mechanisms such as executive functioning through neuroplasticity-enhancing modalities.

[Objectives of the Clinical Trial]

The aim of this clinical investigation was twofold:

To assess the safety of the investigational digital therapeutic (DTx) device when used by children diagnosed with ADHD.

To evaluate the efficacy of the DTx in improving core symptoms of ADHD compared to a sham (placebo) digital intervention.

[Study Design and Methodology] This was a prospective, multi-center, single-blind, randomized controlled confirmatory trial involving two arms: an experimental group receiving the active digital therapeutic intervention and a control group receiving a digital sham.

The investigational DTx is a game-based software intervention designed to train cognitive flexibility, working memory, and inhibitory control - core executive functions associated with ADHD - through repetitive and engaging digital activities.

-Primary Outcomes: ADHD-RS (Investigator-Rated Scale)

-Secondary Outcomes: Additional cognitive and behavioral endpoints further supported the efficacy of the intervention.

* Parent-rated ADHD-RS-IV (Korean ADHD Rating Scale, K-ARS)
* Stroop Color-Word Interference Test (color-word score)
* Advanced Test of Attention (ATA), visual sensitivity score
* CGI-S(Clinical Global Impression-Severity)
* CGI-I(Clinical Global Impression-Improvement)
* CCTT(Children's Color Trails Test)
* K-CPRS(Korean-Conners Parents Rating Scale)
* WCST(Wisconsin Card Sorting Test)
* Changes in Medication Dosage
* Patient-Reported Outcomes

[Safety Evaluation] Safety was assessed throughout the study period by monitoring adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria:
* Children and adolescents aged 6 years or older but under 13 years, both male and female.
* Diagnosed with ADHD according to DSM-5 criteria or ICD-10 diagnosis of ADHD (F90.0).
* K-ARS scores of 18 or higher for females and 22 or higher for males.
* No changes in ADHD medication dosage or regimen within 1 month prior to enrollment (*For those receiving pharmacological treatment with methylphenidate or amphetamine-based products, a washout period of 14 days is required if they wish to participate after discontinuing medication).
* Medically healthy based on medical history and vital signs assessed during screening, without other medical abnormalities.
* Able to use a smartphone or tablet PC that meets specified requirements to operate the mobile application without difficulty.
* Both the subject and their guardian voluntarily agree to participate and provide written informed consent.

Exclusion Criteria:

* Subjects will be excluded if they meet any of the following criteria:
* Presence of any of the following psychiatric symptoms at baseline: chronic tic disorder (requiring medication), Tourette's disorder, or history of major obsessive-compulsive disorder, schizophrenia, bipolar disorder, post-traumatic stress disorder, conduct disorder, or other childhood psychosis (affective disorders are not exclusionary).
* Wechsler Intelligence Scale for Children (WISC) score below 80.
* Presence of congenital genetic disorders.
* Uncontrolled or severe systemic physical illness requiring hospitalization at baseline.
* Suicide attempt within the past 3 months and assessed as high suicide risk by a psychiatrist.
* Initiation or ongoing other cognitive behavioral therapy within the past 3 months (including any CBT for ADHD or other conditions, based on insurance coverage).
* Presence of visual, auditory, or cognitive impairments.
* Any other reasons deemed by the investigator to make the subject unsuitable for participation in the clinical trial.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ADHD-RS (Investigator-Rated Scale) at end of treatment (FAS) | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  The Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS, Investigator-Rated) is a clinician-administered assessment tool based on the DSM-IV diagnostic criteria for ADHD.
  It includes 18 items, with 9 items assessing inattention and 9 items assessing hyperactivity/impulsivity.
  Each item is scored on a 4-point scale (0 = never or rarely, 3 = very often).
  The total score reflects overall ADHD symptom severity, with higher scores indicating greater severity.
  The investigator-rated version is completed by a trained clinician through interviews and behavioral observations, rather than by parents or teachers.

SECONDARY OUTCOMES:
ADHD-RS-IV (Parent-rated, Korean version) | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  The Attention-Deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV, Parent-rated, Korean version) is a standardized rating scale based on the DSM-IV diagnostic criteria for ADHD.
  It consists of 18 items corresponding to the inattention (9 items) and hyperactivity/impulsivity (9 items) symptom domains.
  Parents rate the frequency of each symptom on a 4-point Likert scale ranging from 0 (never or rarely) to 3 (very often).
  The Korean version has been translated and validated for use in Korean populations.
  Higher scores indicate greater severity of ADHD symptoms.
CGI-S(Clinical Global Impression-Severity) | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  The Clinical Global Impression - Severity (CGI-S) scale is a 7-point clinician-rated scale that assesses the clinician's global impression of the patient's current illness severity at the time of evaluation.
  The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  It provides a simple, standardized measure of overall illness severity, independent of specific symptom rating scales.
CGI-I(Clinical Global Impression-Improvement) | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  The Clinical Global Impression - Improvement (CGI-I) scale is a 7-point clinician-rated scale used to assess how much a patient's illness has improved or worsened relative to baseline.
CCTT(Children's Color Trails Test) | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  The Children's Color Trails Test (CCTT) is a neuropsychological assessment tool designed to evaluate cognitive functions in children, particularly:
  * Attention and sustained focus
  * Cognitive flexibility (set-shifting, task-switching)
  * Processing speed
  * Executive functioning
Stroop | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  The Stroop Test (Stroop Color and Word Test) is a widely used neuropsychological assessment designed to measure attention, selective attention, processing speed, and inhibitory control, which are key aspects of executive function.
Changes in Medication Dosage | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  Changes in Medication Dosage refers to any adjustments in the dose of a participant's prescribed ADHD medication during the study period.
Patient-Centered Outcomes | The digital therapy was administered over 4 weeks, including 6-7 visits (2-3 onsite, 4 phone). Screening and Baseline visits could occur on the same day. Final follow-up took place at week 4 post-treatment.
  Satisfaction (10-point)
  Participants will rate their overall satisfaction with the intervention on a 10-point Visual Analog Scale (VAS), with higher scores indicating greater satisfaction.
  Task Difficulty (10-point)
  Participants will rate the perceived difficulty of the tasks on a 10-point VAS, with higher scores indicating greater difficulty.
  Suggestions for Improvement (Open-ended)
  Participants can provide subjective comments or suggestions regarding the intervention.
  Willingness to Pay (Objective)
  Participants will indicate their willingness to pay for the intervention using a structured, objective questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Emotiv, Seoul, gangnam, South Korea

IPD SHARING:
Plan to Share IPD: No